CLINICAL TRIAL: NCT05179447
Title: Randomized Phase III Trial of Molecular Profile-based Versus Standard Recommendations for Adjuvant Therapy for Women With Early Stage Endometrioid Adenocarcinoma
Brief Title: PROfiling Based Endometrial Cancer Adjuvant Therapy
Acronym: PROBEAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Collaborators: Tongji Hospital (Other); Qilu Hospital of Shandong University (Other); Obstetrics & Gynecology Hospital of Fudan University (Other); Sun Yat-sen University (Other); Peking University People's Hospital (Other); Shanghai First Maternity and Infant Hospital (Other); Xiangya Hospital of Central South University (Other); Anhui Provincial Cancer Hospital (Other); Ningbo Women & Children's Hospital (Other); Ningbo No. 1 Hospital (Other)
Responsible Party: Principal Investigator, Wang Xinyu, Clinical Professor, Women's Hospital School Of Medicine Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-20210340-R
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Endometrial Cancer Stage I; Endometrial Cancer Stage II
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Observation; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Molecular profile based treatment (Experimental): Determination of the integrated genomic-pathologic profile to determine adjuvant treatment: observation for POLE-mutated profile; vaginal brachytherapy for intermediate profile; chemo-radiotherapy for p53-abnormal profile.
  Interventions: Radiation: Vaginal brachytherapy; Other: Observation; Combination Product: Chemoradiation therapy
- Radiotherapy (Active Comparator): Adjuvant vaginal brachytherapy for intermediate risk (stage I A with G3 or stage I B with G1-2) and external beam pelvic radiotherapy for high-intermediate risk (stage I B with G3, or stage II) (standard treatment)
  Interventions: Radiation: Vaginal brachytherapy; Radiation: External beam radiotherapy

INTERVENTIONS:
Radiation: Vaginal brachytherapy — Internal radiation of the vaginal vault using a vaginal cylinder. For brachytherapy administered alone it is recommended: suggested dose is either 3 fractions of 7 Gy or 5 fractions of 6 Gy.
  For brachytherapy administered after completion of External beam radiotherapy (EBRT):
  Total dose should aim to be 65 Gy, and suggested dose is 2-3 fractions of 5-6 Gy
Radiation: External beam radiotherapy — External beam pelvic radiotherapy on a linear accelerator, 45-50 Gy in 25-28 out-patients sessions
  Arms: Radiotherapy
Other: Observation — No adjuvant therapy, but active follow-up and quality of life questionnaires as in the groups who have adjuvant treatment
  Arms: Molecular profile based treatment
Combination Product: Chemoradiation therapy — 4 adjuvant cycles carboplatin and paclitaxel followed by External beam pelvic radiotherapy (45-50 Gy )
  Arms: Molecular profile based treatment

SUMMARY:
This is a prospective, multicenter, randomized phase III trial among women with endometrioid adenocarcinoma with high-intermediate and intermediate risk features to investigate the role of integrated genomic-pathologic classification to determine if participants should receive no adjuvant therapy, vaginal brachytherapy, external beam radiotherapy or chemo-radiation therapy based on molecular features as compared to standard radiation therapy.

DETAILED DESCRIPTION:
Adjuvant therapy for women with endometrial cancer has increasingly been tailored to prognostic factors to prevent overtreatment and select those women for adjuvant treatment who will have a clinically relevant reduction of the risk of relapse by the adjuvant treatment. Risk profiles have traditionally been based on clinicopathological factors such as age, stage, grade, Lymph-Vascular Space Invasion (LVSI) and depth of invasion. Newer, both molecular-genetic (the cancer genome atlas subgroups) have become available which are strongly related to outcomes and risk of cancer spread. Based on 2022 National Comprehensive Cancer Network (NCCN) guideline and the ongoing "Portec-4a" trial, this randomized trial using integrated genomic-pathologic classification to assign adjuvant treatment for women with stage I-II high-intermediate and intermediate risk endometrioid adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Surgery consisting of a total abdominal or laparoscopic hysterectomy, bilateral salpingectomy, pelvic lymphadenectomy or sentinel lymph node mapping and dissection, with or without para-aortic lymphadenectomy, oophorectomy
2. Histologically confirmed endometrioid type endometrial carcinoma, International Federation of Gynecology and Obstetrics (FIGO) 2009 stage I, with one of the following combinations of stage and grade:

   Stage I A, grade 3 Stage I B, grade 1 or 2 Stage I B, grade 3 Stage II
3. World Health Organization (WHO)-performance status 0-2
4. Written informed consent

Exclusion Criteria:

1. With residual disease
2. Any other stage and type of endometrial carcinoma
3. Histological types serous carcinoma or clear cell carcinoma (at least 10% if mixed type), or undifferentiated or neuroendocrine carcinoma
4. Uterine sarcoma (including carcinosarcoma)
5. Previous malignancy (except for non-melanomatous skin cancer)
6. Previous pelvic radiotherapy
7. Expected interval between the operation and start of radiotherapy exceeding 8 weeks

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Total recurrence | 3 years
  Vaginal, pelvic or distant recurrence as first failure

SECONDARY OUTCOMES:
Relapse-free survival | 3 years, 5 years
  Relapse-free survival (survival without relapse)
Survival | 3 years, 5 years
  Overall survival (all-cause death)
Adverse events | 3 years, 5 years
  Treatment-related symptoms according to CTCAE v 5.0
Health-related cancer-specific quality of life | 3 years, 5 years
  Quality of Life Core Questionnaire (QLQC-30) - clinically relevant changes on Quality of Life Core Questionnaire-30 functioning scales, general quality of life and general cancer symptoms, quite a bit/very much vs no or mild symptoms
Endometrial cancer related health care costs | 3 years, 5 years
  All hospital based health care costs used with primary treatment or during followup for treatment of adverse events and/or treatment for relapse

OTHER OUTCOMES:
Recurrence (vaginal and total) per risk profile | 3 years, 5 years
  Vaginal, pelvic and distant relapse split by risk profile and compared between the 2 arms

CONTACTS AND LOCATIONS:
Overall Officials: Xinyu Wang, MD, Principal Investigator — Women's Hospital School Of Medicine Zhejiang University
Locations (10):
- China (10):
  - Tongji Hospital, Huazhong University of Science and Technology, Wuhan, Hubei
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Women's Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang
  - Peking University Peoples Hospital, Beijing
  - Xiangya Hospital of Central South University, Changsha
  - Sun Yat-Sen University Cancer Hospital, Guangzhou
  - Ningbo First Hospital, Ningbo
  - Ningbo Women and Children's Hospital, Ningbo
  - Obstetrics & Gynecology Hospital of Fudan University, Shanghai
  - Shanghai First Maternity and Infant Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Concin N, Matias-Guiu X, Vergote I, Cibula D, Mirza MR, Marnitz S, Ledermann J, Bosse T, Chargari C, Fagotti A, Fotopoulou C, Gonzalez Martin A, Lax S, Lorusso D, Marth C, Morice P, Nout RA, O'Donnell D, Querleu D, Raspollini MR, Sehouli J, Sturdza A, Taylor A, Westermann A, Wimberger P, Colombo N, Planchamp F, Creutzberg CL. ESGO/ESTRO/ESP guidelines for the management of patients with endometrial carcinoma. Int J Gynecol Cancer. 2021 Jan;31(1):12-39. doi: 10.1136/ijgc-2020-002230. Epub 2020 Dec 18. PMID 33397713
- [Background] Leon-Castillo A, de Boer SM, Powell ME, Mileshkin LR, Mackay HJ, Leary A, Nijman HW, Singh N, Pollock PM, Bessette P, Fyles A, Haie-Meder C, Smit VTHBM, Edmondson RJ, Putter H, Kitchener HC, Crosbie EJ, de Bruyn M, Nout RA, Horeweg N, Creutzberg CL, Bosse T; TransPORTEC consortium. Molecular Classification of the PORTEC-3 Trial for High-Risk Endometrial Cancer: Impact on Prognosis and Benefit From Adjuvant Therapy. J Clin Oncol. 2020 Oct 10;38(29):3388-3397. doi: 10.1200/JCO.20.00549. Epub 2020 Aug 4. PMID 32749941
- [Background] Wortman BG, Bosse T, Nout RA, Lutgens LCHW, van der Steen-Banasik EM, Westerveld H, van den Berg H, Slot A, De Winter KAJ, Verhoeven-Adema KW, Smit VTHBM, Creutzberg CL; PORTEC Study Group. Molecular-integrated risk profile to determine adjuvant radiotherapy in endometrial cancer: Evaluation of the pilot phase of the PORTEC-4a trial. Gynecol Oncol. 2018 Oct;151(1):69-75. doi: 10.1016/j.ygyno.2018.07.020. Epub 2018 Aug 3. PMID 30078506
- [Background] de Boer SM, Powell ME, Mileshkin L, Katsaros D, Bessette P, Haie-Meder C, Ottevanger PB, Ledermann JA, Khaw P, Colombo A, Fyles A, Baron MH, Jurgenliemk-Schulz IM, Kitchener HC, Nijman HW, Wilson G, Brooks S, Carinelli S, Provencher D, Hanzen C, Lutgens LCHW, Smit VTHBM, Singh N, Do V, D'Amico R, Nout RA, Feeney A, Verhoeven-Adema KW, Putter H, Creutzberg CL; PORTEC study group. Adjuvant chemoradiotherapy versus radiotherapy alone for women with high-risk endometrial cancer (PORTEC-3): final results of an international, open-label, multicentre, randomised, phase 3 trial. Lancet Oncol. 2018 Mar;19(3):295-309. doi: 10.1016/S1470-2045(18)30079-2. Epub 2018 Feb 12. PMID 29449189
- [Background] Leon-Castillo A, Britton H, McConechy MK, McAlpine JN, Nout R, Kommoss S, Brucker SY, Carlson JW, Epstein E, Rau TT, Bosse T, Church DN, Gilks CB. Interpretation of somatic POLE mutations in endometrial carcinoma. J Pathol. 2020 Mar;250(3):323-335. doi: 10.1002/path.5372. Epub 2020 Jan 29. PMID 31829442
- [Derived] Li Y, Zhu C, Xie H, Chen Y, Lv W, Xie X, Wang X. Molecular profile-based recommendations for postoperative adjuvant therapy in early endometrial cancer with high-intermediate or intermediate risk: a Chinese randomized phase III trial (PROBEAT). J Gynecol Oncol. 2023 Mar;34(2):e37. doi: 10.3802/jgo.2023.34.e37. Epub 2023 Jan 10. PMID 36659832